CLINICAL TRIAL: NCT07272590
Title: An Open, Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of QLC5513 in Combination With Epalolimab Tovolimab (QL1706) ± Platinum in Patients With Advanced or Metastatic Malignant Solid Tumors
Brief Title: Study of QLC5513 in Combination With Epalolimab Tovolimab (QL1706) ± Platinum in Patients With Advanced or Metastatic Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLC5513-201
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Solid Tumors
MeSH Terms: interventions — Infusions, Intravenous; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: QLC5513+QL1706 (Experimental)
  Interventions: Drug: QLC5513 IV infusion; Biological: QL1706, IV infusion
- Arm B: QLC5513+QL1706+ platinum (Experimental)
  Interventions: Drug: QLC5513 IV infusion; Biological: QL1706, IV infusion; Drug: platinum, IV infusion

INTERVENTIONS:
Drug: QLC5513 IV infusion — Participants will receive QLC5513 16 mg/kg intravenously on Days1, Day 8 and Day 15 of 28-day cycles.
Biological: QL1706, IV infusion — QL1706 5mg/kg intravenously on Day 1 of 21-day.
Drug: platinum, IV infusion — Cisplatin: 75 mg/m ² or carboplatin：AUC=5 mg/mL/min on Day 1 of 21-day.
  Arms: Arm B: QLC5513+QL1706+ platinum

SUMMARY:
The goal of this Phase Ib/II interventional study is to evaluate the safety, tolerability, pharmacokinetics and efficacy of QLC5513 combined with QL1706± platinum in the treatment of patients with advanced or metastatic malignant solid tumors. This study is divided into two phases: Phase Ib is the combined dose escalation phase, where dose escalation of QLC5513 combined with QL1706± platinum is conducted and RP2D is explored; In the Phase II tumor type expansion study stage, the primary objective is to evaluate the objective response rate (ORR) of QLC5513 combined with QL1706± platinum-based treatment in patients with advanced or metastatic malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Has an eastern cooperative oncology group (ECOG) performance status of 0 to 1.
2. Has adequate organ function.
3. The expected survival period is ≥3 months.
4. Based on the pathological report of the most recent biopsy or other pathological specimens, advanced or metastatic solid tumors confirmed by histology or cytology are not suitable for radical treatments such as surgery and radiotherapy.
5. According to the RECIST v1.1 evaluation criteria, the participants had at least one radiologically measurable lesion.

Exclusion Criteria:

1. Prior treatment with TROP2-targeting agents, ADCs with topoisomerase 1 inhibitor (TOP1i) payloads, or other TOP1i drugs.
2. There was symptomatic central nervous system (CNS) metastasis, leptomeningeal metastasis or spinal cord compression caused by metastasis before the first use of the investigational product.
3. Active, uncontrolled bacterial, fungal or viral infections.
4. Radiotherapy with more than 25% of the bone marrow exposed within 4 weeks prior to the first use of the investigational drug; Local radiotherapy (excluding brain radiotherapy) was performed within two weeks before the first use of the investigational drug.
5. Subjects with a history of a second malignant tumor other than the target indication within 5 years prior to signing the informed consent (excluding cured basal cell skin cancer, superficial bladder cancer, carcinoma in situ of the breast, papillary thyroid carcinoma, etc.).
6. Prior to the first dose of the investigational product, all reversible toxicities from prior anti-tumor therapy (excluding alopecia and pigmentation) have not recovered to ≤ Grade 1 (as assessed by CTCAE v5.0), with the exception that peripheral neuropathy must have not recovered to ≤ Grade 2. History of irAEs from prior immune checkpoint inhibitor treatment that required permanent discontinuation of the immune checkpoint inhibitor.
7. Active autoimmune disease that has required systemic treatment in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD)/maximum administration dose (MAD) and RP2D of QLC5513 combined with QL1706± platinum in patients with advanced solid tumors. | up to 12 months
Number of participants who experience one or more adverse events(AEs). | up to 48 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Objective Response Rate | up to 36 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by investigator.

SECONDARY OUTCOMES:
DOR | up to 48 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by investigator.
PFS | up to 48 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version1.1 (RECIST 1.1). PD is defined as ≥20%increase in the sum of diameters of target lesions. In addition to the relative increase of20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearanceof one or more new lesions is alsoconsidered PD. PFS as assessed by investigator.
OS | up to 60 months
  OS is defined as the time from randomization to death due to any cause.